CLINICAL TRIAL: NCT05978284
Title: A Phase 1/2 Dose Escalation Study of the Tolerability, Safety, Efficacy and Pharmacokinetics of ZG006 in Participants With Small Cell Lung Cancer or Neuroendocrine Carcinoma
Brief Title: Study of ZG006 in Participants With Small Cell Lung Cancer or Neuroendocrine Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZG006-001
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Small Cell Lung Cancer; Neuroendocrine Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Neuroendocrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): During the dose-escalation, an accelerated titration design (ATD) will be utilized for the first two dose groups (0.03mg and 0.1 mg), and the conventional "3+3" dose escalation method will be used for the subsequent dose groups. The entire duration of 28 days after the first dose of ZG006 is defined as the dose-limiting toxicity (DLT).
  Interventions: Biological: ZG006
- Part 2: Dose Expansion (Experimental): Participants will receive the RP2D/MTD identified in Part 1 (dose exploration) of the study.
  Interventions: Biological: ZG006

INTERVENTIONS:
Biological: ZG006 — ZG006 will be administered as an intravenous (IV) infusion.

SUMMARY:
This is a multi-center, open-label, Phase Ⅰ/Ⅱ clinical study of ZG006 for the treatment of participants with small cell lung cancer or neuroendocrine carcinoma who had no standard treatment available, or were intolerant to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form;
* Male or female 18~75 years of age;
* Histologically or cytologically confirmed diagnosis of small cell lung cancer (SCLC), neuroendocrine carcinoma (NEC), who had no standard treatment available, or were intolerant to standard treatments;
* Archival tissue sample or fresh biopsy tissue sample must be available for DLL3 detection;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
* Life expectancy ≥ 3 months;
* Must have evaluable or measurable lesion. For lesions that have received radiation therapy, only after the progression of the lesions, they can be considered evaluable or measurable lesions;
* All adverse events from prior treatment have either returned to baseline or CTCAE 5.0 ≤ Grade 1, except for AEs not constituting a safety risk in the opinions of the investigators, e.g. alopecia, hypothyroidism which can be treated with a hormone replacement, etc.;
* Female and Male patients must agree to use a reliable form of contraception during the study treatment period and for at least 6 months after the last dose of the study drug.

Exclusion Criteria:

* Patients having received any of the following treatments:

Anti-DLL3 and anti-CD3 drugs (including investigational drugs); Chemotherapy, biotherapy, endocrine therapy (except for hormone replacement), and biological targeted medicines ≤ 4 weeks before the study entry. Local palliative radiotherapy and a small molecule targeted therapy ≤ 2 weeks (or 5 half-lives, whichever is longer) before the study entry; Systemic immunosuppressive medications, such as corticosteroid (doses > 10 mg/day prednisone or equivalent dose) within 14 days prior to the study entry; Use of any vaccines against viral infections (COVID-19, influenza, varicella, etc.) within 4 weeks of study entry;

* Received any blood transfusion, EPO, G-CSF, albumin infusion and renal replacement therapy within 14 days prior to study entry.
* The main organ function meets any of the following criteria within 7 days prior to study entry; Hematological function: ANC < 1.5×10^9/L, PLT < 75×10^9/L, Hemoglobin (Hb) < 100 g/L; Hepatic function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 3×ULN, ALT and AST ≥ 5×ULN for liver metastases patients; Total bilirubin (TBIL) ≥ 1.5×ULN; albumin < 30g/L; Creatinine clearance (Cockcroft-Gault formula) < 50 mL/min; INR > 1.5 or APTT > 1.5×ULN;
* Medical history, computed tomography (CT) or magnetic resonance imaging (MRI) results indicate the existence of central nervous system (CNS) metastases; Note: Not applicable to the following conditions: subjects with stable CNS metastases;
* Uncontrollable third cavity effusion (e.g. a large amount of pleural effusion, ascites, or pericardial effusion, etc.) requiring repeated drainage, which was judged by the investigator to be unsuitable for study;
* Any other malignancy within 5 years (other than radically removed and has not recurred tumors including basal cell skin carcinoma, squamous cell skin carcinoma, superficial bladder cancer, localized prostate cancer, cervical cancer and other cancer in situ, etc.);
* Severe cardiac-cerebral vascular disease, including but not limited to:

Acute myocardial infarction, unstable angina, stroke, or received coronary angioplasty or stent implantation within 6 months before study entry; New York Heart Association functional class II to IV congestive heart failure or left ventricular ejection fraction (LVEF) < 50% or the lower limit of normal; Uncontrollable hypertension (even though the best treatment is used but systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg).

QTc (F) interval prolonged in electrocardiography during the screening baseline period (> 480 ms)

* History of autoimmune disease, including but not limited to systemic lupus erythematosus, nephritis, psoriasis, rheumatoid arthritis, inflammatory bowel disease, autoimmune hepatitis (except for the following: type I diabetes mellitus, skin diseases that do not require systemic treatment (such as vitiligo), controllable celiac disease, and childhood asthma that completely resolved in adulthood without intervention);
* Active infection (such as acute bacterial infection, tuberculosis, active hepatitis B/C, active syphilis, or active human immunodeficiency virus infection). Active hepatitis B is defined as: hepatitis B virus DNA titer > 10000 copies/mL or 2000 IU/mL; active hepatitis C is defined as: a positive hepatitis C antibody and HCV viral load above the limit of quantification; active human immunodeficiency virus infection is defined as: antibody positive;
* Active neurologic paraneoplastic syndrome;
* Interstitial lung disease or non-infectious pneumonitis (other than radiation-induced pneumonia);
* Having received prior allogeneic stem cell transplantation or solid organ transplantation;
* Known allergy to other mAbs or any antibody excipients; the history of a severe allergic reaction, anaphylactoid or other hypersensitivity reactions to humanized antibodies or fusion proteins;
* Known history of diagnosed neurological or mental disorders, for example, epilepsy, dementia, etc.;
* A female who is pregnant or nursing;
* Patients were deemed unsuitable for participating in the study by the investigator for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicity (DLT) | Up to 28 days
  An event is considered to be a DLT if the event occurs within the first 28 days of treatment and meets the dose-limiting toxicity criteria
Maximum Tolerated Dose (MTD) of ZG006 | Up to approximately 1 year
Determine the Recommended Phase 2 Dose (RP2D) | Up to approximately 1 year
Number of participants with adverse events (AEs) | Up to approximately 2 year
  The types and frequencies of adverse events (AEs) evaluated according to the National Cancer Institute Common Terminology Criteria for adverse events (NCI-CTCAE) version 5.0
Number of participants with serious adverse events (SAEs) | Up to approximately 2 year
Incidence of abnormal laboratory results | Up to approximately 2 year
  Abnormal laboratory results of safety concerns such as ALT, AST, Cr and BUN, et al according to NCI-CTCAE 5.0 classification.
Changes of ECGs from baselines | Up to approximately 2 year
  Changes of ECGs from baselines, such as QT interval

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 2 year
  ORR is defined as the percentage of participants achieving a confirmed complete response (CR) or partial response (PR) based on RECIST 1.1 criteria.
Duration of response (DOR) | Up to approximately 2 year
  DOR is defined as the time from first evidence of response (CR or PR per RECIST 1.1) to earlier date of disease progression or death due to any cause
disease control rate (DCR) | Up to approximately 2 year
Maximum plasma concentration (Cmax) of ZG006 | Baseline and up to approximately 1 year
Time to peak concentration (Tmax) | Up to approximately 1 year
AUC from time zero to the last quantifiable concentration after dosing (AUC[0-t]) of ZG006 | Up to approximately 1 year
Terminal phase half-life (t1/2) of ZG006 | Up to approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Qiming Wang, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China